CLINICAL TRIAL: NCT00077792
Title: A Randomized, Double-Blind, Double-Dummy , Parallel Group, Multinational, Clinical Study to Evaluate the Efficacy and Safety of Enoxaparin Versus Unfractionated Heparin in Patients With Acute ST-Segment Elevation Myocardial Infarction Receiving Fibrinolytic Therapy
Brief Title: Enoxaparin and Thrombolysis Reperfusion for Acute Myocardial Infarction Treatment Thrombolysis in Myocardial Infarction - Study 25 (ExTRACT-TIMI25)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC6147; XRP4563B/3001
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Myocardial Infarction; Acute ST-Segment Elevation
Keywords: Receiving fibrinolytic therapy
MeSH Terms: conditions — Myocardial Infarction | interventions — enoxaparin sodium

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Enoxaparin sodium (XRP4563)

SUMMARY:
The primary objective of the study is to determine whether enoxaparin compared to unfractionated heparin will reduce the composite endpoint of all-cause mortality and non-fatal myocardial re-infarction within 30 days after randomization in patients with acute ST-segment elevation myocardial infarction who are eligible to receive fibrinolytic therapy

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with ST-segment elevation acute myocardial infarction meeting all of the following criteria:

* Male or non-pregnant female greater than or equal to 18 years of age (depending on local regulations, minimal age can vary between 18 and 21 years)
* Onset of prolonged (greater than or equal to 20 min) ischemic symptoms at rest less than or equal to 6 hours prior to randomization
* ST-segment elevation of 0.1 mV in 2 or more limb leads, or 0.2 mV in two (2) or more contiguous precordial leads, or left bundle-branch block
* Planned reperfusion therapy with streptokinase, tenecteplase, alteplase or reteplase
* Written informed consent will be obtained

EXCLUSION CRITERIA:

Cardiovascular

* Evidence of cardiogenic shock at randomization
* Acute pericarditis
* History or symptoms suggestive of aortic dissection
* MI precipitated by obvious provoking factors such as arrhythmia, infection, severe anemia, hyperthyroidism, cocaine, or amphetamine

Hemorrhagic Risk

* Any minor head trauma or any other trauma occurring after the index acute myocardial infarction
* Active or recent (< 3 months) bleeding including gastrointestinal bleeding, known presence of occult blood in the stool, or gross hematuria.
* Any history of bleeding diathesis, coagulopathy, platelet disorder, or thrombocytopenia
* Any single reliable recording of systolic blood pressure >180 mm Hg and/or diastolic blood pressure >110 mm Hg prior to randomization
* Any history of stroke or transient ischemic attack; any history of hemorrhagic cerebrovascular disease
* Any known structural damage or other pathologic process involving the central nervous system
* Any head trauma within 6 months prior to randomization
* Major surgery (including CABG), any ophthalmologic surgery, or non-cutaneous biopsy, or substantial trauma within 3 months prior to randomization
* Traumatic or prolonged cardiopulmonary resuscitation (> 2 minutes) within 2 weeks prior to randomization
* Puncture of a non-compressible vessel (artery or vein) within the 24 hours prior to randomization
* Acute peptic ulcer disease within 3 months prior to randomization

Prior or Concomitant Pharmacologic Therapy

* Administration of abciximab (ReoPro), within the previous 7 days or eptifibatide (Integrilin), or tirofiban (Aggrastat) within the previous 24 hours prior to randomization
* Current therapy with oral anticoagulants, or an International Normalized Ratio of >1.5
* Administration of a low molecular weight heparin within 8 hours prior to randomization.
* Known hypersensitivity to low molecular weight heparins, unfractionated heparin or heparin-like products; allergy to pork or pork products
* Known hypersensitivity and/or contra-indication(s) to fibrinolytic drugs (streptokinase, tenecteplase, alteplase and reteplase)

General

* Known platelet count <100,000 cells/microL or history of heparin-induced thrombocytopenia
* Known clinically significant anemia (Hemoglobin <10 g/dL which is < 6.2 mmol/L)
* Known renal insufficiency with serum creatinine >220 mmol/L (2.5 mg/dL) for men and >175 mmol/L (2.0 mg/dL) for women when assessed prior to baseline examination.
* Advanced neoplastic or other life-threatening disease with a life expectancy of <12 months
* Pregnancy or parturition within the last 90 days or currently breast feeding
* Women of childbearing potential except if post-menopausal, surgically sterile or using accepted method(s) of birth control or having a negative pregnancy test.
* Treatment with other investigational agents in the last 30 days before study entry or previous enrollment in ExTRACT-TIMI 25
* History of drug or alcohol abuse
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study
* Any patient unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and who are unlikely to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20506 (Actual)
Dates: Start 2002-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality and non-fatal myocardial re-infarction

SECONDARY OUTCOMES:
Composite of all-cause mortality, non-fatal myocardial re-infarction, and myocardial ischemia leading to urgent revascularization and non-fatal disabling stroke

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (48):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- sanofi-aventis administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Minsk, Belarus
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shangaï, China
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi- Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Dublin, Ireland
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Amman, Jordan
- Sanofi-Aventis Administrative Office, Riga, Latvia
- Sanofi-Aventis Administrative Office, Beirut, Lebanon
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- Sanofi-aventis adminsitrative office, Guildford Surrey, United Kingdom
- Sanofi-Aventis Administrative Office, Montevideo, Uruguay

REFERENCES:
- [Result] Antman EM, Morrow DA, McCabe CH, Murphy SA, Ruda M, Sadowski Z, Budaj A, Lopez-Sendon JL, Guneri S, Jiang F, White HD, Fox KA, Braunwald E; ExTRACT-TIMI 25 Investigators. Enoxaparin versus unfractionated heparin with fibrinolysis for ST-elevation myocardial infarction. N Engl J Med. 2006 Apr 6;354(14):1477-88. doi: 10.1056/NEJMoa060898. Epub 2006 Mar 14. PMID 16537665
- [Derived] Morrow DA, Antman EM, Fox KA, White HD, Giugliano R, Murphy SA, McCabe CH, Braunwald E; ExTRACT-TIMI 25 Investigators. One-year outcomes after a strategy using enoxaparin vs. unfractionated heparin in patients undergoing fibrinolysis for ST-segment elevation myocardial infarction: 1-year results of the ExTRACT-TIMI 25 trial. Eur Heart J. 2010 Sep;31(17):2097-102. doi: 10.1093/eurheartj/ehq098. Epub 2010 Apr 17. PMID 20400762